CLINICAL TRIAL: NCT06287528
Title: A Phase I Trial of CD19-targeted Chimeric Antigen Receptor (CAR) T Cells That Constitutively Secrete Interleukin 18 (19-28z/IL-18) in Patients With Relapsed or Refractory (R/R) Acute Lymphoblastic Leukemia (ALL)
Brief Title: A Study of 19-28z/IL-18 in People With Acute Lymphoblastic Leukemia (ALL)
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 23-307
Record Dates: First submitted 2024-02-23; First posted 2024-03-01 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Philadelphia-Negative ALL; Philadelphia-Positive ALL; Relapsed ALL, Adult; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia (ALL); Refractory Acute Lymphoid Leukemia in Relapse
Keywords: Philadelphia-Negative ALL; Philadelphia-Positive ALL; Philadelphia chromosome negative (Ph-negative) B-ALL; Philadelphia chromosome positive (Ph+ positive) B-ALL; Relapsed ALL, Adult; Refractory Acute Lymphoblastic Leukemia; Refractory Acute Lymphoblastic Leukemia (ALL); Refractory Acute Lymphoid Leukemia in Relapse; 19-28z/IL-18; 23-307; Memorial Sloan Kettering Cancer Center
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Dose Level 1 (Experimental): 0.5x106 CAR-T cell/kg without lymphodepleting chemotherapy (LDC)
  Interventions: Biological: 19-28z/IL-18 CAR T cells
- Dose Level 2 (Experimental): 0.5x106 cells/kg with lymphodepleting chemotherapy (LDC)
  Interventions: Biological: 19-28z/IL-18 CAR T cells
- Dose Level 3 (Experimental): 1x106 cells/kg with lymphodepleting chemotherapy (LDC)
  Interventions: Biological: 19-28z/IL-18 CAR T cells

INTERVENTIONS:
Biological: 19-28z/IL-18 CAR T cells — 19-28z/IL-18 CAR T cells are an investigational new drug (IND) for the treatment of R/R B-ALL

SUMMARY:
Participants will have a sample of their white blood cells, called T cells, collected using a procedure called leukapheresis. The collected T cells will be sent to a laboratory to be changed (modified) to become 19-28z/IL-18, the CAR T-cell therapy that participants will receive during the study. Making the participants' study therapy will take about 2-4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have R/R ALL meeting one of the following criteria:
* For Philadelphia chromosome (Ph) negative B-ALL: Refractory or relapsed disease to at least 1 prior multiagent systemic chemotherapy regimen that included both induction and consolidation therapy
* For Philadelphia chromosome (Ph) positive B-ALL: patients must have exhibited persistent or progressive disease following at least 1 prior second- or third-generation tyrosine kinase inhibitor
* Signed informed consent form (ICF) prior to any study procedures
* Age: The first 3 patients enrolled into the study will be ≥ 17 years of age at time of enrollment. If a DLT is observed, the additional 3 patients in this cohort will also be ≥ 17 years of age. Additional patients will be ≥12 years of age at time of enrollment.
* Documentation of CD19 positivity on leukemia blasts if prior anti-CD19 treatment
* History of prior allogeneic hematopoietic stem cell transplant (HSCT) is allowed if ≥3 months from time of enrollment and no evidence of acute or chronic graft versus host disease (GVHD) within 4 weeks prior to enrollment
* Donor lymphocyte infusions (DLI) permitted if ≥4 weeks prior to leukapheresis
* History of secondary CNS or meningeal involvement allowed if:

  * cannot be the only site of disease
  * absence of neurologic symptoms, such as: seizures, stroke-like deficits, altered mental status, aphasia, or psychosis
* Adequate organ function at time of screening, including:

  * ALT or AST ≤5x ULN and total bilirubin ≤2 (or ≤3 if history of Gilbert's syndrome or leukemic infiltration of the liver)
  * Serum creatinine <2.0mg/100mL
  * SaO2 ≥92% on room air
  * Left ventricular ejection fraction (LVEF) ≥50% within 1 month of screening
* ECOG performance status 0-1 or Lansky performance status ≥ 60 for patients < 16 years old
* Prior CD19-targeted therapies (including CD19 CAR-T cell and CD19 bispecific T-cell engagers) are allowed including anti-CD19 CAR T therapy, as long as CD19 positivity is confirmed on most recent bone marrow, blood or tumor biopsy

Exclusion Criteria:

* Concurrent active malignancy excluding: nonmelanoma skin cancer or localized solid tumor that has undergone definitive therapy and with low risk of recurrence, e.g., prostate, breast
* Burkitt's leukemia or lymphoma or CML in lymphoid blast crisis
* Radiologically detected or symptomatic CNS disease or CNS 3 disease (i.e., presence of ≥5/µL WBCs in CSF). Subjects with adequately treated CNS leukemia are eligible.
* The following medications are excluded:

  * Steroids: Therapeutic doses of corticosteroids (greater than 10mg daily of prednisone or its equivalent) within 7 days of leukapheresis or 72 hours prior to CAR T cell infusion.
  * Chemotherapy: Systemic chemotherapy should be stopped one week prior to leukapheresis or starting CAR T cell infusion or lymphodepleting chemotherapy. Hydroxyurea for cytoreduction can be administered up to 72 hours before leukapheresis or CAR T cell infusion.
* History of class III-IV New York Heart Association (NYHA) heart failure, cardiac angioplasty or stenting, myocardial infarction, unstable angina, or other clinically significant cardiac condition within 6 months of screening
* Patients with history of significant autoimmune disease and/or inflammatory condition affecting the CNS are ineligible
* Systemic treatment for GVHD within 4 weeks prior to enrollment
* Patients with known severe autoimmune disease (e.g., Crohn's, rheumatoid arthritis, or lupus) that in the investigator's opinion has high likelihood of requiring systemic immune suppressive medications
* Patients with HIV infection
* Patients with active hepatitis B infection (as manifested by either detectable hepatitis B virus DNA by PCR and/or positivity for hepatitis B surface antigen)
* Patients with active hepatitis C infection (as manifested by detectable hepatitis C virus RNA by PCR)
* Patients with uncontrolled systemic fungal, bacterial, viral or other infection including COVID-19 at time of leukapheresis or at time of CAR T cell infusion.
* Other uncontrolled medical or psychological conditions as well as social or logistical issues that may interfere with compliance with the protocol, as determined by the investigator
* Treatment with live, attenuated vaccine <4 weeks prior to leukapheresis
* Pregnant or lactating/breastfeeding women

Min Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2024-02-23 (Actual); Primary Completion 2028-02-23 (Estimated); Study Completion 2028-02-23 (Estimated)

PRIMARY OUTCOMES:
Toxicity as determined by CTCAE, version 5.0 | 4 weeks
  The primary objective is to determine the safety of 19-28z/IL18 CAR T cells in patients with R/R ALL. Toxicity will be graded on a scale of 1 to 5 as described by the NCI Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Jae Park, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (7):
- United States (7):
  - Memorial Sloan Kettering at Basking Ridge (Limited Protocol Activities), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Limited Protocol Activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Limited Protocol Activities), Montvale, New Jersey
  - Memorial Sloan Kettering Cancer Suffolk-Commack (Limited Protocol Activities), Commack, New York
  - Memorial Sloan Kettering Westchester (Limited Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (Limited Protocol Activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org